CLINICAL TRIAL: NCT02924038
Title: Pilot Randomized Neo-adjuvant Evaluation of Agonist Anti-CD27 Monoclonal Antibody Varlilumab on Immunologic Activities of IMA950 Vaccine Plus Poly-ICLC in Patients With WHO Grade II Low-Grade Glioma (LGG)
Brief Title: A Study of Varlilumab and IMA950 Vaccine Plus Poly-ICLC in Patients With WHO Grade II Low-Grade Glioma (LGG)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Industry sponsor decision
Sponsor: Nicholas Butowski (Other)
Collaborators: Celldex Therapeutics (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Nicholas Butowski, MD, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15108; NCI-2017-01369 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); 5R21CA233856-02 (NIH)
Record Dates: First submitted 2016-05-12; First posted 2016-10-05 (Estimated); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Glioma; Malignant Glioma; Astrocytoma, Grade II; Oligodendroglioma; Glioma, Astrocytic; Oligoastrocytoma, Mixed
Keywords: low-grade glioma; glioma; immunotherapy; vaccine; WHO grade II
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma; Lymphoma, Follicular | interventions — IMA950; poly ICLC; varlilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IMA950/poly-ICLC subcutaneous (subQ) + Varlilumab IV (Experimental): IMA950 4.96mg and poly-ICLC 1.4mg administered as one formulation subcutaneously followed immediately by a Varlilumab 3mg/kg infusion (intravenously) -23±2 days (about 3 weeks) before the date of scheduled standard-of-care surgery to remove the WHO grade II glioma. Patients will continue receiving IMA950/poly-ICLC subcutaneous injections every week leading up to surgery (Days -16±2, -9±2 and 24-48 hours prior to scheduled surgery) and every 3 weeks after surgery (Weeks A1, A4, A7, A10, A13, A16, A19, A22; defining Week A1 as the first post-surgery vaccine). After surgery, patients will continue receiving a Varlilumab infusion every 6 weeks immediately following the IMA950/poly-ICLC injection (Weeks A1, A7, A13, and A19).
  Interventions: Biological: IMA950; Biological: poly-ICLC; Biological: Varlilumab
- IMA950/poly-ICLC subQ only (Experimental): IMA950 4.96mg and poly-ICLC 1.4mg administered as one formulation subcutaneously every week leading up to standard-of-care surgery to remove the WHO grade II glioma (Days -23±2, -16±2, -9±2 and 24-48 hours prior to scheduled surgery) and every three weeks after surgery (Weeks A1, A4, A7, A10, A13, A16, A19, A22; defining Week A1 as the first post-surgery vaccine). Patients will not receive Varlilumab.
  Interventions: Biological: IMA950; Biological: poly-ICLC

INTERVENTIONS:
Biological: IMA950 — IMA950 vaccine
  Other Names: IMA950 peptides
Biological: poly-ICLC — poly-ICLC vaccine
  Other Names: Hiltonol
Biological: Varlilumab — Intravenous solution
  Other Names: CDX-1127
  Arms: IMA950/poly-ICLC subcutaneous (subQ) + Varlilumab IV

SUMMARY:
This is a pilot, randomized, two arm neoadjuvant vaccine study in human leukocyte antigen-A2 positive (HLA-A2+) adults with World Health Organization (WHO) grade II glioma, for which surgical resection of the tumor is clinically indicated. Co-primary objectives are to determine: 1) the safety of the novel combination of subcutaneously administered IMA950 peptides and poly-ICLC (Hiltonol) and i.v. administered CDX-1127 (Varlilumab) in the neoadjuvant approach; and 2) whether addition of i.v. CDX-1127 (Varlilumab) increases the response rate and magnitude of CD4+ and CD8+ T-cell responses against the IMA950 peptides in post-vaccine peripheral blood mononuclear cell (PBMC) samples obtained from participating patients.

DETAILED DESCRIPTION:
Low-grade gliomas (LGG), the most common of which are pilocytic astrocytomas, diffuse astrocytomas, and oligodendrogliomas are a diverse family of central nervous system (CNS) neoplasms that occur in children and adults. Based on data from the American Cancer Society and Central Brain Tumor Registry of the United States (CBRTUS), approximately 1,800 LGG were diagnosed in 2006, thus representing approximately 10% of newly diagnosed primary brain tumors in the United States. Pilocytic astrocytomas (WHO grade I) are the most common brain tumor in children 5 to 19 years of age. Diffuse astrocytomas and oligodendrogliomas are all considered WHO grade II low grade gliomas (LGG) and are more common in adults. Pilocytic astrocytomas are generally well circumscribed histologically and radiographically and amenable to cure with gross total resection. In contrast, the diffuse astrocytomas and oligodendrogliomas are more infiltrative and less amenable to complete resection. From a molecular genetics standpoint, the most common alterations in LGG are Isocitrate dehydrogenase 1 (IDH1) mutations and mutations in the tumor suppressor gene tumor protein 53 (TP53), located on chromosome 17, the gene product of which is a multi-functional protein involved in the regulation of cell growth, cell death (apoptosis), and transcription. Additionally, several molecular factors are of favorable prognostic significance, particularly the presence of 1p/19q co-deletion and isocitrate dehydrogenase (IDH) mutations.

WHO grade II LGGs are at risk to undergo malignant transformation into more aggressive and lethal WHO grade III or IV high-grade glioma (HGG). Even with a combination of available therapeutic modalities (i.e., surgery, radiation therapy (RT), chemotherapy), the invasive growth and resistance to therapy exhibited by these tumors results in recurrence and death in most patients. Although postoperative RT in LGG significantly improves 5-year progression-free survival (PFS), it does not prolong overall survival (OS) compared with delayed RT given at the time of progression. Early results from a randomized trial of radiation therapy plus procarbazine, lomustine, and vincristine (PCV) chemotherapy for supratentorial adult LGG (RTOG 9802) demonstrated improved PFS in patients receiving PCV plus RT compared RT alone. Nonetheless, PCV is considerably toxic and currently not widely used for management of glioma patients. Although chemotherapy with temozolomide (TMZ) is currently being investigated in LGG patients, it is unknown whether it confers improved OS in these patients. Further, our recent study has indicated that 6 of 10 LGG cases treated with TMZ progressed to HGG with markedly increased exome mutations and, more worrisome, driver mutations in the retinoblastoma tumor suppressor (RB) and Protein kinase B (AKT)-Mechanistic target of rapamycin (mTOR) pathways, with predominant C>T/G>A transitions at CpC and CpT dinucleotides, strongly suggesting a signature of TMZ-induced mutagenesis; this study also showed that in 43% of cases, at least half of the mutations in the initial tumor were undetected at recurrence, while IDH mutations were the only type of mutations that persisted in the initial and recurrent tumors. These data suggests the possibility that treatment of LGG patients with TMZ may enhance oncogenic mutations and genetic elusiveness of LGG, therefore calling for development of safer and effective therapeutic modalities such as vaccines.

Taken together, LGG are considered a premalignant condition for HGG, such that novel interventions to prevent malignant transformation need to be evaluated in patients with LGG. Immunotherapeutic modalities, such as vaccines, may offer a safe and effective option for these patients due to the slower growth rate of LGG (in contrast with HGG), which should allow sufficient time for multiple immunizations and hence high levels of anti-glioma immunity. Because patients with LGGs are generally not as immuno-compromised as patients with HGG, they may also exhibit greater immunological response to and benefit from the vaccines. Further, the generally mild toxicity of vaccines may improve quality of life compared with chemotherapy or RT.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >= 18 years old.
* Pathological criteria - Participants must have a newly diagnosed or recurrent WHO grade II astrocytoma, oligoastrocytoma or oligodendroglioma that has been histologically confirmed by prior biopsy or surgical resection. If the pathological diagnosis ws made outside of University of California, San Francisco (UCSF), the pathology must be reviewed and confirmed at UCSF.
* Patients must be positive for HLA-A2 based on flow-cytometry or genotyping
* Before enrollment, patients must show non-enhancing T2-FLAIR lesions lesions that are amenable to surgical resection. Surgical resection of at least 0.3 grams of tumor is expected to ensure adequate evaluation of the study endpoints
* Prior radiation therapy (RT) after the initial diagnosis will be allowed but there must be at least 6 months from the completion of RT (or radiosurgery) to signed informed consent.
* Prior chemotherapy and any systemic molecularly targeted anti-tumor therapy will be allowed, and there must be at least 28 days from the last temodar chemotherapy, 42 days for nitrosourea; at least 14 days from the last dose for chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity.
* Patients must have a Karnofsky performance status (KPS) of >= 70%.
* Off or low dose (<= 4 mg/day by Decadron) corticosteroid at least two weeks before the first pre-surgical vaccine
* Adequate organ function within 28 days of study registration including: 1) Adequate bone marrow reserve: absolute neutrophil (segmented and bands) count (ANC) >=1.0 x 10^9/L, absolute lymphocyte count >=4.0 x 10^8/L, platelets >=100 x 10^9/L; hemoglobin >=8 g/dL; 2) Hepatic: - Total bilirubin <= 1.5 x upper limit of normal (ULN) and Serum glutamic pyruvic transaminase(SGPT)/ (alanine aminotransferase (ALT)) <=2.5 x upper limit of normal (ULN), and 3) Renal: Normal serum creatinine or creatinine clearance >=60 ml/min/1.73 m^2
* Must be free of systemic infection. Subjects with active infections (whether or not they require antibiotic therapy) may be eligible after complete resolution of the infection. Subjects on antibiotic therapy must be off antibiotics for at least 7 days before beginning treatment.
* Sexually active females of child bearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device (IUD), surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of the vaccination period. Sexually active males must agree to use barrier contraceptive for the duration of the vaccination period.
* Women of child-bearing potential and men must agree to use adequate contraception (ex. Hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation (until one month after the last vaccine) since the effects of the current regimen on the developing human fetus are unknown. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Patient must sign an informed consent document indicating that they are aware of the investigational nature of this study, which includes an authorization for the release of their protected health information

Exclusion Criteria:

* Presence of gliomatosis cerebri, cranial or spinal leptomeningeal metastatic disease
* Presence of T1 Gadolinium (Gd)-enhancing lesions (on MRI) suggestive of high-grade glioma
* Pathological diagnosis for the resected tumor demonstrates transformation to higher grade (i.e. WHO grade III or IV) gliomas. If a patient is diagnosed as HGG upon resection after receiving the pre-surgical treatment, the patient will be withdrawn from the study and considered for therapeutic options for HGG (trials for HGG or standard of care). The tumor tissue of such a case would be brought to the lab before the pathological diagnosis is made; and thus would be processed before the lab is informed of the final HGG diagnosis. Because HGG tissue may still reflect the vaccine effects, we will evaluate the tumor tissue to help us develop future approaches for HGG.
* Pregnant women are excluded from this study because IMA950 and poly-ICLC are drugs with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with IMA950 plus poly-ICLC (IMA950-poly-ICLC hereafter) vaccine, breastfeeding should be discontinued if the mother is treated with IMA950- poly-ICLC vaccine
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection (e.g. active or chronic hepatitis B and C), symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* History or current status of immune system abnormalities such as hyperimmunity (e.g., autoimmune diseases) that needed to be treated by systemic therapy, such as immuno-suppressants and hypoimmunity (e.g., myelodysplastic disorders, marrow failures, AIDS, transplant immunosuppression).
* Any isolated laboratory abnormality suggestive of a serious autoimmune disease (e.g. hypothyroidism): Antinuclear antibody, thyroid-stimulating hormone (TSH), free thyroxine (FT4), rheumatoid factor
* Any condition that could potentially alter immune function (AIDS, multiple sclerosis, diabetes, renal failure)
* Receiving ongoing treatment with immunosuppressive drugs or dexamethasone > 4mg
* Use of any of the following concurrent treatment or medications:

  * radiation therapy
  * chemotherapy
  * interferon (e.g. Intron-A)
  * allergy desensitization injections
  * growth factors (e.g. Procrit, Aranesp, Neulasta)
  * Interleukins (e.g. Proleukin)
  * any investigational therapeutic medication
* Prior cancer diagnosis except the following:

  * squamous cell cancer of the skin without known metastasis
  * basal cell cancer of the skin without known metastasis
  * carcinoma in situ of the breast (DCIS or LCIS)
  * carcinoma in situ of the cervix
* Any other acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with trial participation or trial drug administration or could interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into the trial.
* Participants with known addiction to any drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hideho Okada, MD, PhD, Principal Investigator — University of California, San Francisco; Nicholas Butowski, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saijo A, Ogino H, Butowski NA, Tedesco MR, Gibson D, Watchmaker PB, Okada K, Wang AS, Shai A, Salazar AM, Molinaro AM, Rabbitt JE, Shahin M, Perry A, Clarke JL, Taylor JW, Daras M, Oberheim Bush NA, Hervey-Jumper SL, Phillips JJ, Chang SM, Hilf N, Mayer-Mokler A, Keler T, Berger MS, Okada H. A combinatory vaccine with IMA950 plus varlilumab promotes effector memory T-cell differentiation in the peripheral blood of patients with low-grade gliomas. Neuro Oncol. 2024 Feb 2;26(2):335-347. doi: 10.1093/neuonc/noad185. PMID 37758193

RESULTS

PARTICIPANT FLOW:
Groups:
- IMA950/Poly-ICLC Subcutaneous (subQ) + Varlilumab IV: IMA950 4.96mg and poly-ICLC 1.4mg administered as one formulation subcutaneously followed immediately by a Varlilumab 3mg/kg infusion (intravenously) -23±2 days (about 3 weeks) before the date of scheduled standard-of-care surgery to remove the World Health Organization (WHO) grade II glioma. Patients will continue receiving IMA950/poly-ICLC subcutaneous injections every week leading up to surgery (Days -16±2, -9±2 and 24-48 hours prior to scheduled surgery) and every 3 weeks after surgery (Weeks A1, A4, A7, A10, A13, A16, A19, A22; defining Week A1 as the first post-surgery vaccine). After surgery, patients will continue receiving a Varlilumab infusion every 6 weeks immediately following the IMA950/poly-ICLC injection (Weeks A1, A7, A13, and A19).
Period: Overall Study
Arm/Group | IMA950/Poly-ICLC Subcutaneous (subQ) + Varlilumab IV | IMA950/Poly-ICLC subQ Only
Started | 8 | 6
Included in Biological Analysis | 6 | 5
Completed | 6 | 4
Not Completed | 2 | 2
Not completed — Excluded from post-surgery vaccines due to high-grade diagnosis of resected tumor | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IMA950/Poly-ICLC Subcutaneous (subQ) + Varlilumab IV | IMA950/Poly-ICLC subQ Only | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Customized [Count of Participants; unit: Participants]
  20-29 years old | 2 | 1 | 3
  30-39 years old | 1 | 1 | 2
  40-49 years old | 3 | 4 | 7
  50-59 years old | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 5 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Experiencing Regimen Limiting Toxicity (RLT)
Description: The proportion of participants experiencing and RLT defined as an adverse event judged to be possibly, probably or definitely associated with treatment that requires participants to be taken off study and no further injections will be given will be reported.
Time Frame: up to 2 years
Measure: Number; unit: proportion of participants
Arm/Group | IMA950/Poly-ICLC Subcutaneous (subQ) + Varlilumab IV | IMA950/Poly-ICLC subQ Only
Number analyzed (Participants) | 8 | 6
proportion of participants | 0 | 0

2. Primary Outcome: Mean Percentage of CD8+ T-cell Responses in Pre- and Post-vaccine Peripheral Blood Mononuclear Cells (PBMC)
Description: The expansion of IMA950-reactive CD8+ T cell frequencies over post-vaccine periods was assessed by calculating the mean percentage of total IMA950 tetramer-positive CD8+ T cell per available post-vaccine time point. CD8+ T-cell response to the IMA950-epitope is defined to be positive when the percentage of tetramer-positive CD8+ T cells showed a four-fold or higher increase within at least one-time point in the post-vaccine phase relative to the corresponding percentage at the pre-vaccine.
Time Frame: Up to 2 years
Measure: Mean (Standard Deviation); unit: percentage of T cell responses
Arm/Group | IMA950/Poly-ICLC Subcutaneous (subQ) + Varlilumab IV | IMA950/Poly-ICLC subQ Only
Number analyzed (Participants) | 6 | 5
percentage of T cell responses
  Pre-Vaccine Cluster 3 Effector CD8 | 4.5 (4.2) | 7.3 (3.6)
  Post-Vaccine Cluster 3 Effector CD8 | 12.5 (8.0) | 13.3 (8.3)
  Pre-vaccine Cluster 8 Effector memory | 2.2 (1.0) | 2.7 (2.2)
  Post-vaccine Cluster 8 Effector memory | 5.9 (2.3) | 4.5 (4.6)

3. Primary Outcome: Mean Percentage of CD4+ T-cell Responses in Pre- and Post-vaccine PBMC
Description: The expansion of IMA950-reactive CD4+ T cell frequencies over post-vaccine periods was assessed by calculating the mean percentage of total IMA950 tetramer-positive CD4+ T cell per available post-vaccine time point. CD4+ T-cell response to the IMA950-epitope is defined to be positive when the percentage of tetramer-positive CD4+ T cells showed a four-fold or higher increase within at least one-time point in the post-vaccine phase relative to the corresponding percentage at the pre-vaccine.
Time Frame: Up to 2 years
Population: Data not collected.
Arm/Group | IMA950/Poly-ICLC Subcutaneous (subQ) + Varlilumab IV | IMA950/Poly-ICLC subQ Only
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | IMA950/Poly-ICLC Subcutaneous (subQ) + Varlilumab IV | IMA950/Poly-ICLC subQ Only
All-Cause Mortality (participants affected / at risk) | 1/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/6
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMA950/Poly-ICLC Subcutaneous (subQ) + Varlilumab IV (N=8) | IMA950/Poly-ICLC subQ Only (N=6)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMA950/Poly-ICLC Subcutaneous (subQ) + Varlilumab IV (N=8) | IMA950/Poly-ICLC subQ Only (N=6)
Injection site reaction (General disorders) | 8 (135) | 6 (56)
Fatigue (General disorders) | 4 (7) | 6 (26)
Flu like symptoms (General disorders) | 4 (36) | 2 (2)
Fever (General disorders) | 1 (4) | 3 (3)
Pain (General disorders) | 2 (3) | 1 (2)
Chills (General disorders) | 0 (0) | 1 (1)
Edema face (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (6) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (12) | 4 (22)
Nervous system disorders - Other, specify (Nervous system disorders) | 4 (5) | 3 (4)
Seizure (Nervous system disorders) | 1 (1) | 3 (4)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 1 (2) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 6 (7) | 2 (8)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 4 (5) | 1 (2)
Lymphocyte count decreased (Investigations) | 6 (24) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (4) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (4) | 1 (1)
White blood cell decreased (Investigations) | 3 (14) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (13) | 3 (9)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (5) | 1 (7)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (6) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (6) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (7) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 3 (8) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 1 (1)
Blurred vision (Eye disorders) | 1 (2) | 0 (0)
Retinal vascular disorder (Eye disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (4)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment was closed earlier than expected due to industry sponsor's prioritization of other programs, the termination of Varliumab development, and Coronavirus disease of 2019 (COVID-19) related challenges during the period of enrollment. Appropriate reagents were not available for the CD4+ outcome measure. Due to the small number of participants, the biological/immunological evaluations are insufficiently powered to provide meaningful statistical significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT02924038/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT02924038/ICF_001.pdf